CLINICAL TRIAL: NCT03353376
Title: Group Versus Individual Care in Patients With Long Standing Type 1 and Type 2 Diabetes: Non Inferiority in a One Year Prospective Study in a Tertiary Diabetes Clinic
Brief Title: Group Versus Individual Care in Diabetes Clinic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rabin Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: JSMG-01
Record Dates: First submitted 2017-11-02; First posted 2017-11-27 (Actual); Last update posted 2017-11-27 (Actual); Status verified 2017-10

CONDITIONS: Diabetes Mellitus; Group Meetings
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group care with empowerment model (Experimental): 4 group visits a year according to empowerment model in a tertiary diabetes clinic
  Interventions: Behavioral: group care with Empowerment model
- individual usual care (Active Comparator): individual visits according to disponibility in the diabetes clinic and needs of the patients
  Interventions: Behavioral: group care with Empowerment model

INTERVENTIONS:
Behavioral: group care with Empowerment model — Patients with type 2 and type 1 diabetes were followed in a tertiary outpatient clinic with group appointment

SUMMARY:
In this prospective, randomized, non blinded, one center (University hospital) trial, 60 patients (28 with type 1 and 32 with type 2 diabetes) with a mean duration of diabetes of 22.5 ± 11.7 years were randomly assigned to group (6 patients per group) or individual usual care for one year. Primary end-point included change in Hba1c and visits to out-patients clinics, secondary endpoint included change in body mass index, blood pressure levels, waist circumference, non HDL Cholesterol, diabetes related and quality of life questionnaires and hospitalizations.

DETAILED DESCRIPTION:
in the intervention arm patients attended 4 preplanned group visits in the study year and the empowerment model was used in the group care visits.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 1 or type 2 diabetes
* Fluency in Hebrew
* Attendance at least for the second time at the diabetes clinic
* Follow up of at least one year by a general practitioner
* Willingness to participate in the study and to give informed consent.

Exclusion Criteria:

* Uncontrolled psychiatric diseases
* Active cancer
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-09-13 (Actual); Primary Completion 2014-01-02 (Actual); Study Completion 2014-01-02 (Actual)

PRIMARY OUTCOMES:
change in in Hba1c levels | one year from date of randomization
  Collection of data at start and after one year

SECONDARY OUTCOMES:
change in scores of diabetes specific questionnaire | one year from date of randomization
  Collection of data at start and end of study from electronic files
change in BMI in kg/m2 | one year from date of randomization
  Collection of data (weight in kg, height in meter) at start and end of study from electronic files
change in non HDL Cholesterol | one year from date of randomization
  Collection of data at start and end of study from electronic files

OTHER OUTCOMES:
change in number of outpatients visits | one year from date of randomization
  Collection of data at start and after one year
change in number in hospital admission | one year from date of randomization
  Collection of data at start and end of study from electronic files

CONTACTS AND LOCATIONS:
Overall Officials: Noa Naftali, MA, Study Chair — Rabin Medical Center